CLINICAL TRIAL: NCT05423808
Title: Streamlined Geriatric and Oncological Evaluation Based on IC Technology for Holistic Patient-oriented Healthcare Management for Older Multimorbid Patients. TWOBE Study
Brief Title: Geriatric and Oncological Evaluation With Technology for Holistic Healthcare Management for Older Multimorbid Patients.
Acronym: GerOnTe-TWOBE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: important delays in digital health tool development made the timelines unfeasible within the project
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Bordeaux (Other); Diakonessenhuis, Utrecht (Other); University of Milan (Other); University College Dublin (Other); Oslo University Hospital (Other); International Society of Geriatric Oncology (Other); Dublin City University (Other); Universitair Ziekenhuis Brussel (Other); General Hospital Groeninge (Other); AZ Sint-Jan AV (Other); Catharina Ziekenhuis Eindhoven (Other); Reinier de Graaf Groep (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: s66300
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-12

CONDITIONS: Geriatrics; Medical Oncology; Critical Pathways; Digital Technology
Keywords: Geriatrics; Oncology; Patient-centred care; Technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: stepped wedge randomized controlled trial (cross-over type)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will be part of a renewed care pathway supported by digital tools.
  Interventions: Other: Health Professional Consortium; Device: Holis Dashboard - Holis Patient App
- Control group (No Intervention): Patients in the control group will receive standard of care, specific to the hospital where the patient is being treated.

INTERVENTIONS:
Other: Health Professional Consortium — In the intervention group, the renewed, patient-centred care pathway will be coordinated by the Advanced Practice Nurse (APN) and will be supported by digital technology. The intervention aims to increase the involvement of the patient in the treatment decision process, to provide comprehensive care through the quarterly meeting of all professionals involved in the care of the patient during a Health Professional Consortium (HPC) and to support patient empowerment by supporting self-management by using digital tools.
  Arms: Intervention group
Device: Holis Dashboard - Holis Patient App — In the intervention group, the renewed, patient-centred care pathway will be coordinated by the Advanced Practice Nurse (APN) and will be supported by digital technology. The intervention aims to increase the involvement of the patient in the treatment decision process, to provide comprehensive care through the quarterly meeting of all professionals involved in the care of the patient during a Health Professional Consortium (HPC) and to support patient empowerment by supporting self-management by using digital tools.
  Arms: Intervention group

SUMMARY:
The GerOnTe TWOBE study aims to evaluate the effectiveness of the GerOnTe intervention, consisting of a renewed, patient-centred, care pathway coordinated by an APN and supported by a Health Professional Consortium and IC Technology, compared to the current standard of care in the eight different Belgian and Dutch hospitals.

DETAILED DESCRIPTION:
The GerOnTe TWOBE study aims to evaluate the effectiveness of the GerOnTe intervention, consisting of a renewed, patient-centred, care pathway coordinated by an APN and supported by a Health Professional Consortium and IC Technology, compared to the current standard of care in the eight different Belgian and Dutch hospitals. The GerOnTe project consists of two identical trials in two different European geographical areas, FRONE in France and TWOBE in Belgium and the Netherlands. The goal of two identical trials is to take into account the role of health care contexts in the implementation, effectiveness and efficiency of the GerOnTe intervention. A stepped wedge randomized controlled trial, where the randomized clusters will be participating hospitals, will be conducted in eight academic and general hospitals in total with a follow-up at 3, 6, 9 and 12 months after study inclusion. Patients will be recruited in all participating hospitals in the period between the cancer diagnosis and the treatment decision.

ELIGIBILITY:
General inclusion criteria:

1. Age ≥ 70 years old,
2. New or progressive cancer (breast, lung, colorectal, prostate) fulfilling the tumour specific inclusion criteria,
3. Estimated life expectancy greater than 6 months,
4. At least one moderate/severe multimorbidity inclusion criteria other than current cancer (separate list),
5. Patients must be willing and able to comply with study procedures,
6. Voluntarily signed and dated written informed consents prior to any study specific procedure,
7. QLQ-C30 Quality of Life Questionnaire fully completed at baseline, before inclusion.

Tumour specific inclusion criteria:

8. Specific inclusion criteria for breast cancer: 8.1. Non-metastatic breast cancer (M0):

* No prior treatment for the current breast cancer.
* All 3 criteria required:

  * Clinical staging: cT2-3-4 Nany, or cTany N1-2-3,
  * The cancer specialist considers* surgery,
  * The cancer specialist considers* radiotherapy and/or chemotherapy. 8.2. Metastatic breast cancer (M1): Both criteria required:
* The cancer specialist considers* chemotherapy or PARP-inhibitors or mTOR-inhibitors / PIK3CA inhibitors; Previous endocrine therapy +/- CDK4/6 inhibitors is allowed,
* The patient received maximum 1 prior line of chemotherapy for metastatic disease.

  *'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

  9. Specific inclusion criteria for colorectal cancer: 9.1. Non-metastatic colorectal cancer (M0):
* No prior therapy for the current tumour in the recruiting hospital.
* At least one of the 3 criteria required:

  - The cancer specialist considers* surgery,

  - The cancer specialist considers* radiotherapy,

  - The cancer specialist considers* chemotherapy. 9.2. Metastatic colorectal cancer (M1):
* The cancer specialist considers* first line systemic therapy and/or radiotherapy (+/- surgery). No previous chemotherapy allowed except adjuvant/perioperative chemotherapy stopped for more than 12 months.

  *'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

  10. Specific inclusion criteria for lung cancer: 10.1. Non-metastatic lung cancer (M0):
* No prior therapy for the current tumour in the recruiting hospital.
* At least one of the 3 criteria required:

  * The cancer specialist considers* surgery (patients considered for treatment with percutaneous thermoablation alone are not eligible),
  * The cancer specialist considers* radiotherapy (except SBRT),
  * The cancer specialist considers* systemic therapy. Possible systemic therapies are chemotherapy and/or immune therapy and/or targeted therapy. Patients only considered* for monotherapy with anti-EGFR TKI or somatostatin analog are not eligible.

10.2. Metastatic lung cancer (M1):

* The cancer specialist considers* first or second line systemic therapy. Possible systemic therapies are chemotherapy and/or immune therapy and/or targeted therapy. Patients only considered* for monotherapy with anti-EGFR TKI or somatostatin analog are not eligible.

  *'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

  11. Specific inclusion criteria for prostate cancer: 11.1. Non-metastatic prostate cancer (M0): one of the following:
* First diagnosis M0 prostate cancer (no therapy received yet for prostate cancer): at least one of the 2 criteria required:

  - The cancer specialist considers* radiotherapy,
  * The cancer specialist considers* hormone therapy (ADT +/- combination Abiraterone and Prednisone).
* Salvage treatment M0 prostate cancer (received prior surgery at least 6 months before):

  * The cancer specialist considers* radiotherapy (+/- ADT).
* Non-metastatic castration resistant prostate cancer:

  * The cancer specialist considers* treatment intensification (ADT + Enzalutamide or Apalutamide or Darolutamide).

11.2. Metastatic prostate cancer (M1): • The cancer specialist considers* treatment with Abiraterone or Enzalutamide or Apalutamide, or Docetaxel or Cabazitaxel or PARP-inhibitors or Lutetium PSMA.

*'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

Exclusion criteria:

1. Mental illness/cognitive impairment that limits ability to provide consent or complete trial procedures.
2. Participating to an interventional clinical trial with a non-registered anticancer drug or to another geriatric intervention trial.
3. Patients and caregivers are unable or unwilling to use ICT-devices (tablet, computer, smartphone) or the Internet according to protocol.
4. Patient already included in this study.

Separate list of severe morbidity criteria:

General

1. Two or more unscheduled comorbidity related hospitalisations in the past year (not related to index cancer).
2. Having received out-patient care from two more specialties in the past year (not related to index cancer).

   Cardiac
3. Any prior symptomatic myocardial infarction.
4. Any past valve replacement, percutaneous coronary intervention), percutaneous transluminal coronary angioplasty) or coronary artery bypass graft.
5. Congestive heart failure under follow-up by a cardiologist.
6. Chronic exertional angina.
7. Regular use of anti-anginal medication.
8. Left ventricular hypertrophy.
9. Dyspnoea or activity restriction secondary to cardiac status.
10. One or more admissions to hospital for cardiac reasons in past year.

    Vascular
11. Previous vascular intervention.
12. Symptomatic atherosclerotic/peripheral vascular disease.

    Venous
13. Any history of pulmonary embolism.
14. Use of coumadin/warfarin, heparin, DOAC or NOAC with indication venous disease.

    Hypertension
15. Need of three or more types of blood pressure medication.

    Haematopoetic
16. Any chronic hematologic disease.
17. Haemoglobin: <10 g/dL (6.0 mmol/l) (not related to index cancer).

    Endocrine
18. Insulin dependence.
19. Diabetes-related complications (retinopathy, neuropathy, nephropathy, coronary artery disease or peripheral arterial disease).
20. Poorly controlled diabetes mellitus or diabetic coma in the past year.
21. Requires adrenal hormone replacement.

    Pulmonary
22. Dyspnoea at rest.
23. Limited activities secondary to pulmonary status.
24. Requires oral steroids for lung disease.
25. One or more admissions to hospital for pulmonary reasons in past year.
26. Two or more hospitalisations for pneumonia in past five years.

    Renal
27. eGFR < 30 ml/min.

    Hepatobilary
28. Chronic hepatitis.
29. Cirrhosis.
30. Portal hypertension with moderate symptoms.
31. Compensated liver failure.
32. Clinical or lab evidence of biliary obstruction (not related to index cancer).
33. Acute or chronic pancreatitis or hepatitis in past 5 years.

    Stomach/intestine
34. Recent ulcers (<6 months) or any history of ulcers requiring hospitalisation.
35. Any history of inflammatory bowel disease.
36. Any swallowing disorder or dysphagia.
37. Chronic diarrhoea (not related to index cancer).
38. Bowel impaction in the past year (not related to index cancer).
39. Status post bowel obstruction (not related to index cancer).
40. Ostomy/stoma in situ (not related to index cancer).

    Nutrition and weight
41. Weight loss more than 6 kg in past six months.
42. Weight loss more than 3 kg in past 1 month.
43. Significantly decreased food intake.
44. Body mass index < 19 kg/m2.
45. Body mass index > 38 kg/m2.

    Neurologic
46. Status post cerebrovascular accident (CVA) with at least mild residual dysfunction.
47. Any past central nervous system neurosurgical procedure.
48. Neurodegenerative disease including Parkinson's disease, parkinsonism, multiple sclerosis, myasthenia gravis etc.).
49. Requires daily meds for chronic headaches or headaches that regularly interfere with daily activities.

    Sensory
50. Partially or functionally blind, unable to read newsprint.
51. Functional deafness or conversational hearing impaired despite hearing aid.
52. Laryngectomy.

    Mobility
53. Requires a walking aid/wheelchair.
54. Difficulties in activities of daily living secondary to mobility impairment.
55. Difficulty walking >100m without resting.
56. Requires steroids or immunosuppressant medication for arthritic condition or connective tissue disease.
57. Prior or current symptomatic vertebral compression fractures from osteoporosis.

    Psychiatric
58. Active substance abuse with social, behavioural or medical complications.
59. History of schizophrenia or another psychotic disorder.
60. Requires daily antipsychotic medication.
61. Current usage of daily anti-anxiety medication.
62. Currently meets DSM criteria for major depression or bipolar disorder.
63. One or more episodes of major depression in the past 10 years.
64. Any previous psychiatric hospitalisation.

    Cognition/Delirium
65. One or more prior deliriums in the past 10 years.
66. Cognitive impairment that does not inhibit patient to provide informed consent and understand study procedures.

    Previous cancer
67. Another type of cancer than the index cancer with at least one of the following criteria:

    * Required chemotherapy or radiation therapy in the past 5 years,
    * Non-curable and/or metastatic cancer.

    Instrumental Activities of Daily Living (IADL)
68. Care dependent in one or more aspects of the following instrumental activities of daily living (preparing meals, walking outside alone, managing medication).

    Social
69. Patients has no or very limited support system or informal caregivers.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL): EORTC QLQ-C30 | QoL at 6 months after study inclusion
  Quality of Life assessed by the EORTC QLQ-C30 (version 3.0) questionnaire. HRQOL evaluation was performed using the European Organization for Research and Treatment Quality of Life Questionnaire core 30 (EORTC QLQ-C30) Global Health Status Scale (GHS).
  Three derived scores of the QLQ-C30 questionnaire are considered as primary endpoints:
  * Normalized global health status score of the QLQ-C30 (version 3.0) (score 0-100),
  * Normalized score of the physical functioning scale of the QLQ-C30 (version 3.0) (score 0-100),
  * Normalized score of the emotional functioning scale of the QLQ-C30 (version 3.0) (score 0-100).
  A high score for a functional scale represents a high / healthy level of functioning.
  A high score for the global health status / QoL represents a high QoL.

SECONDARY OUTCOMES:
Quality of Life (QoL): EORTC QLQ-C30 | QoL at 3, 9 and 12 months after study inclusion
  HRQOL evaluation was performed using EORTC QLQ-C30 Global Health Status Scale (GHS) and Quality of Life Questionnaire Elderly Cander Patients 14 (EORTC QLQ-ELD14) Global Health Status Scale (GHS).
  * Normalized scores of global health status, physical functioning scale and emotional functioning scale of the QLQ-C30 (version 3.0) (score 0-100).
  * Normalized scores of the QLQ-C30 symptom scales/items (score 0-100).
  * Scores of QLQ-ELD14 scales/items (score 0-100).
  A high score for the global health status / QoL in QLQ-C30 represents a high QoL.
  A high score for a symptom scale / item represents a high level of symptomatology / problems.
  High scores in QLQ-ELD14 indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose, and high burden of illness.
Overall survival | at 12 months after study inclusion
  Survival as the length of time from the start of treatment and death from any cause.
Progression-free survival | at 12 months after study inclusion
  Progression-free survival (PFS) defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first.
Patient autonomy (1) | At baseline, 3, 6, 9 and 12 months after study inclusion
  Dependence score measured by Activities of Daily Living (ADL). The ADL scale includes six items (bathing, dressing, toileting, transferring, continence and feeding), with a score for each item scores ranging from one (able to perform the activity) to four (unable to perform the activity) (range: 6-24).
Patient autonomy (2) | At 6 and 12 months after study inclusion
  Proportion of patients living at home (range: 0-100%). The higher the percentage, the more patients live at home.
Patient autonomy (3) | At baseline, 3, 6, 9 and 12 months after study inclusion
  Number of completed chair stands in 30 seconds measured by the Chair Stand Test. Participants stand up repeatedly from a chair for 30 seconds.
Patient autonomy (4) | At baseline, 3, 6, 9 and 12 months after study inclusion
  The overall level of fitness or frailty of the older patients will be assessed by the 9-point Clinical Frailty Scale (CFS) (score: 1-9).
  The higher the score, the less fit or more frail the older person is.
Patient autonomy (5) | At baseline, 3, 6, 9 and 12 months after study inclusion
  The ECOG Performance Status Scale (ECOG-PS) describes a patient's level of functioning in terms of their ability to care for themself, daily and physical ability (score: 0-5).
  The higher the score, the less active the older person is.
Weight evolution | At baseline, 3, 6, 9 and 12 months after study inclusion
  The weight of a person (in kilograms) measured with a scale.
Patient anxiety | At baseline, 3, 6, 9 and 12 months after study inclusion
  Patient anxiety measured by the Hospital Anxiety and Depression Scale (HADS). The 14 questions can be answered by a 4-point Likert scale (0-3). The odd questions (1, 3, 5, 7, 9, 11, 13) refer to fear (score: 0-21).
  The higher a person scores on this questionnaire, the more complaints of anxiety he/she experiences.
Patient institutionalisation | At baseline, 6 and 12 months after study inclusion
  Proportion of patients institutionalised (see definition) (range: 0-100%). Definition: Institutionalisation means that a patient moves permanently to an institution among which are considered retirement houses.
Patient unscheduled hospitalisations | During 12 months after study inclusion
  Proportion of patients with at leas one unscheduled hospitalisation and number of unscheduled hospitalisations per patient (see definition) (range: 0-100%).
  Definition: Unscheduled hospitalisation includes any hospitalisation which has not been previously planned because of an unscheduled event (severe adverse event, complication of treatment, decompensation of morbidity) whatever it is linked or not to the emergency room.
Cost-effectiveness and cost-utility evaluation (1) | During 12 months after study inclusion
  Life years gained (LYG) in the cost per life years gained (CEA) derived from a clinical metric (overall survival/progression-free survival).
Cost-effectiveness and cost-utility evaluation (2) | At baseline, 3, 6, 9 and 12 months after study inclusion
  Quality-adjusted life years (QALYs) in the cost per QALY gained (CUA) calculated using utility assessed through normalised scores of EQ-5D-5L questionnaire. It includes the 5-level questions covering five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 5-digit code for EQ-5D-5L, which reflects how good or bad a health state is according to the preferences of the general population of a country/region (score: 11111-55555 (or 99999 for missing data)).
Cost-effectiveness and cost-utility evaluation (3) | During 12 months after study inclusion
  Total amount resulting from all direct (medical or non-medical) and indirect costs related to disease and care, collected during the 12 months of patient follow-up.
Caregiver burden | At baseline, 3, 6, 9 and 12 months after study inclusion
  Total burden of the caregiver in health, psychological well-being, finances, social life and relationship with the patient will be obtained using the Zarit Burden Interview (ZBI) by adding the scores across all 22 items. Each question is scored on a 5-point scale (score: 0-88).
  The higher the score, the heavier the caregiver burden.
Patient reported overall experience | At 6 and 12 months after study inclusion
  Patient experience of person-centred coordinated care measured through the Person-Centred Coordinated Care Experience Questionnaire (P3CEQ) - 11 items in 5 domains: information and communication processes, care planning, transitions, goals and outcomes and decision making.
Patient, physician and health-care-professionals-reported overall satisfaction with the IC technology of the GerOnTe intervention | At 6 and 12 months after study inclusion
  Patient satisfaction and usability of mHealth application within the GerOnTe intervention will be evaluated by using the score derived from the 21-items mHealth App Usability Questionnaire (MAUQ) for standalone mHealth Apps (Patient version).
  Physician and health-professional satisfaction and usability of mHealth application within the GerOnTe intervention will be evaluated by using the score derived from the adjusted version designed for health care providers of the mHealth App Usability Questionnaire (MAUQ) for standalone mHealth Apps (Provider version), consisted of 18 items.
GerOnTe patient-centred system implementation and usage (1) | At 6 and 12 months after study inclusion
  Number of connections to the Holis Patient App.
GerOnTe patient-centred system implementation and usage (2) | At 6 and 12 months after study inclusion
  Frequency of connections to the Holis Patient App.
GerOnTe patient-centred system implementation and usage (3) | At 6 and 12 months after study inclusion
  Duration of logins and activities with the Holis Patient App,
GerOnTe patient-centred system implementation and usage (4) | At 6 and 12 months after study inclusion
  Number of web-based meetings with Advanced Practice Nurse by site.
GerOnTe patient-centred system implementation and usage (5) | At 6 and 12 months after study inclusion
  Number of Advance Practice Nurse (APN) consultations by site (and by patient).
GerOnTe patient-centred system implementation and usage (6) | At 6 and 12 months after study inclusion
  Number of Patient Reported Outcome Measures (PROM's) dashboards completed by patient (Holis Patient App).
GerOnTe patient-centred system implementation and usage | At 6 and 12 months after study inclusion
  Number of health professional meetings (Multidisciplinary Tumour Boards (MTB) or other morbidities treatment decision) involving complete dashboards analysis by site.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, prof. dr., Principal Investigator — Coordinator multidisciplinary breast centre (MBC)
Locations (1):
- UZ Gasthuisberg Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamaker ME, Wildiers H, Ardito V, Arsandaux J, Barthod-Malat A, Davies P, Degol L, Ferrara L, Fourrier C, Kenis C, Kret M, Lalet C, Pelissier SM, O'Hanlon S, Rostoft S, Seghers N, Saillour-Glenisson F, Staines A, Schwimmer C, Thevenet V, Wallet C, Soubeyran P. Study protocol for two stepped-wedge interventional trials evaluating the effects of holistic information technology-based patient-oriented management in older multimorbid patients with cancer: The GERONTE trials. J Geriatr Oncol. 2024 May;15(4):101761. doi: 10.1016/j.jgo.2024.101761. Epub 2024 Apr 5. PMID 38581958